CLINICAL TRIAL: NCT07030361
Title: Innovative Dialaysis Suit for Hemodialysis Patients Effect of Fluid Restriction on Compliance and Level of Empowerment: Randomise Controlled Trials
Brief Title: Intradıalytıc Weıght Control In Hemodıalysıs Patıents
Acronym: DialysisSuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Türkan Çalışkan, asist proff, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BalikesirUniversity HealtScien; 222S306 (Other Grant/Funding Number: TÜBİTAK)
Record Dates: First submitted 2025-04-17; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fluid Overload
Keywords: FluidControl; Compliance; Empowerment; İnnovation; DialysisSuit;
MeSH Terms: conditions — Edema; Patient Compliance; Empowerment | interventions — Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Intervention Model Description: Research data were collected in 3 stages: pretest (Z0), posttest (Z1) and follow-up test (Z2).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- suits group (Active Comparator): Dialysis suit group was dressed in dialysis suit and given fluid control training
  Interventions: Behavioral: suit group
- 2 training group (Placebo Comparator): Fluid control training was given to the traininig group
  Interventions: Behavioral: training group
- control group (Other): Control group received no intervention, clinical care
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: suit group — elbise giydirme ve video izletme uygulaması
  Arms: suits group
Behavioral: training group — video izletme uygulaması
  Arms: 2 training group
Behavioral: control group — rutin hemş bakımı uygulaması, herhangi bir müdahale yok
  Arms: control group

SUMMARY:
The aim of this observational study is to determine the effect of a dialysis gown designed according to the empowerment model on changes in weight control behaviors among gown group patients during the intradialytic period. The main question it seeks to answer is:

• Is the dialysis gown effective in helping gown group patients control their fluid intake during the intradialytic period?

DETAILED DESCRIPTION:
In this study, researchers designed a study to compare whether the behavior of controlling excessive fluid intake during the intradialytic period was better in the group of patients wearing dialysis garments designed according to the empowerment model than in the education and control groups. For this randomized controlled study, patients were divided into three groups. The patients were named the garment group, the education group, and the control group. In the study design, patients underwent garment application and education application. In the garment application, the amount of excess fluid removed by ultrafiltration during that dialysis session was placed in the pockets of the serum dialysis garment, and patients were asked to walk in a 10-meter walking test area. In the education application, a video-based education program designed to teach fluid compliance behavior was implemented. Patients were asked to watch this video education program for an average of half an hour at the beginning of each session.

Patients in the garment group were dressed in dialysis garments and shown the educational video. Patients in the education group were only shown the fluid compliance video. No intervention specific to the study was performed on patients in the control group. All patients continued to receive the normal follow-up and care protocol required for hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Turkish-speaking
* Turkish-understanding
* Older than 18 years of age
* Without communication barriers such as visual and hearing impairment
* Non-hypotensive and non-anemic patients
* With an intradialytic weight of 2-5 liters
* Receiving hemodialysis treatment for more than three months and outpatients

Exclusion Criteria:

* Patients who had previously received fluid restriction compliance training
* Who refused to participate in the study
* Who had undergone surgery within the last six weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
intradialytic fluid balance | 8 weeks
  weight gained during the intradialytic period

CONTACTS AND LOCATIONS:
Overall Officials: Alper Azak, Asist Prof, Principal Investigator — balikesir
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the product used in the research has not yet entered the production phaset

REFERENCES:
- See also: national thesis center — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp